CLINICAL TRIAL: NCT05016596
Title: Postprandial Lipids in IBS and Nutritional Treatment
Acronym: PLINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Ministry of Economic Affairs (Unknown); Givaudan France Naturals (Industry); Nexira (Industry); Wecare (Other); Roquette Freres (Industry); Ingredion Incorporated (Industry); Ingredia S.A. (Industry); Darling (Unknown); Winclove Probiotics B.V. (Industry); Bioiberica (Industry)
Responsible Party: Principal Investigator, Diederik Esser, Clinical Trial Coordinator, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL75915.041.21
Record Dates: First submitted 2021-07-27; First posted 2021-08-23 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Acacia gum
  Interventions: Dietary Supplement: placebo
- turmeric (Experimental): Turmeric supplement
  Interventions: Dietary Supplement: turmeric

INTERVENTIONS:
Dietary Supplement: turmeric — Turmeric supplement
  Arms: turmeric
Dietary Supplement: placebo — Placebo
  Arms: placebo

SUMMARY:
Irritable Bowel Syndrome (IBS) is a disease that affects a large number of people. Adequate treatment is difficult, partially due to the heterogeneity of the patients and the complicated pathology in which not all mechanisms are understood. Based on literature and in vitro screening within the public private IBSQUtrition consortium project, a turmeric supplement was selected for in vivo validation of its potential beneficial effects on fat-induced intestinal barrier disruption as measured with LPS translocation in IBS patients with a diarrhea-predominant subtype (IBS-D).

The primary objective of this study is to determine the effect of turmeric supplementation on LPS translocation in IBS-D patients after a high-fat challenge. The secondary objective of this study is to determine the effect of turmeric supplementation on gastrointestinal complaints and LPS-related biomarkers in IBS-D patients after a high-fat challenge.

In this double-blind, randomized, placebo-controlled cross-over trial 20 adult (18-70 yrs) IBS-D patients will be included.

Study participants have to invest about 16 hours of their time in this study. They will visit the research facility three times. The risks for participation are very small if not negligible. Consumption of high amounts of saturated fat may cause some gastro-intestinal discomfort. Blood sampling will be performed via a cannula and the insertion can be a bit painful and may cause a bruise. The amount of blood that is drawn from participants is relatively small and within acceptable limits.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients that meet the Rome IV criteria + additional criteria specific for the diarrhea-predominant subtype, based on the most frequent self-reported stool types using the Bristol stool chart
* Male and female adults, aged 18-70 years;
* Having a Body Mass Index (BMI) between 18.5 and 30 kg/m2;
* Willing to keep a stable dietary pattern throughout the study.

Exclusion Criteria:

* Having a disease that may interfere with the outcomes of this study, such as a known autonomic disorder, inflammatory bowel disease, coeliac disease, cancer, dialysis patients, chronic kidney failure, depression or hypothyroidism.
* History of intestinal surgery (excluding appendectomy or cholecystectomy) or endometriosis.
* Use of medication that can interfere with the study outcomes, including codeine and antibiotics, as judged by the medical supervisor.
* Use of anticoagulants (as curcumin has inhibitory effects on platelet aggregation).
* Use of prebiotics and/or probiotics (should be stopped 4 weeks before the start of the study) and infrequent use of other supplements dedicated to bowel function improvements.
* Having swallowing problems with pills/capsules.
* Having a cow's milk allergy or other food allergies.
* If applicable: currently pregnant or breastfeeding, or intending to become pregnant during the study.
* Participation in another clinical trial at the same time.
* Student or employee working at Food, Health and Consumer Research from Food and Biobased Research, or Department of Human Nutrition & Health, Wageningen University.
* Alcohol intake ≥ 14 (women) or ≥ 28 (men) glasses of alcoholic beverages per week.
* Smoking and abuse of illicit drugs, soft drugs, and/or nitrous oxide.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
LPS_B | Baseline
  LPS in venous blood samples collected at baseline
LBP_1 | 1 hour post ingestion
  LBP in venous blood samples collected after high-fat shake consumption.
LPS_2 | 2 hours post ingestion
  LPS in venous blood samples collected after high-fat shake consumption.
LPS_3 | 3 hours post ingestion
  LPS in venous blood samples collected after high-fat shake consumption.
LPS_4 | 4 hours post ingestion
  LPS in venous blood samples collected after high-fat shake consumption.
LPS_5 | 5 hours post ingestion
  LPS in venous blood samples collected after high-fat shake consumption.

SECONDARY OUTCOMES:
ApoB48_B | Baseline
  ApoB48 at baseline
LPB_B | Baseline
  LPB at baseline
sCD14_B | Baseline
  sCD14 at baseline
ApoB48_1 | 1 hour post ingestion
  ApoB48 after high-fat shake consumption
LPB_1 | 1 hour post ingestion
  LPB after high-fat shake consumption
sCD14_1 | 1 hour post ingestion
  sCD14 after high-fat shake consumption
ApoB48_2 | 2 hours post ingestion
  ApoB48 after high-fat shake consumption
LPB_2 | 2 hours post ingestion
  LPB after high-fat shake consumption
sCD14_2 | 2 hours post ingestion
  sCD14 after high-fat shake consumption
ApoB48_3 | 3 hours post ingestion
  ApoB48 after high-fat shake consumption
LPB_3 | 3 hours post ingestion
  LPB after high-fat shake consumption
sCD14_3 | 3 hours post ingestion
  sCD14 after high-fat shake consumption
ApoB48_4 | 4 hours post ingestion
  ApoB48 after high-fat shake consumption
LPB_4 | 4 hours post ingestion
  LPB after high-fat shake consumption
sCD14_4 | 4 hours post ingestion
  sCD14 after high-fat shake consumption
ApoB48_5 | 5 hours post ingestion
  ApoB48 after high-fat shake consumption
LPB_5 | 5 hours post ingestion
  LPB after high-fat shake consumption
sCD14_5 | 5 hours post ingestion
  sCD14 after high-fat shake consumption

OTHER OUTCOMES:
Age | Baseline
  Age
BMI | Baseline
  BMI
Gender | Baseline
  Gender
GI complaints | Baseline
  GI complaints
IBS-related complaints (IBS-SSS) | Baseline
  Severity of IBS-related complaints (IBS-SSS), single score
Stool frequency-3 | -72hr
  Stool frequency on test day -3
Stool frequency-2 | -48hr
  Stool frequency on test day -2
Stool frequency-1 | -24hr
  Stool frequency on test day -1
Stool frequency-T | Testday (0hr)
  Stool frequency on test day
Stool frequency+1 | 24hr
  Stool frequency on test day +1
Stool frequency+2 | 48hr
  Stool frequency on test day +2
Stool consistency-3 | -72hr
  Stool consistency (Bristol stool chart) on test day -3
Stool consistency-2 | -48hr
  Stool consistency (Bristol stool chart) on test day -2
Stool consistency-1 | -24hr
  Stool consistency (Bristol stool chart) on test day -1
Stool consistency-T | Testday (0hr)
  Stool consistency (Bristol stool chart) on test day
Stool consistency+1 | 24hr
  Stool consistency (Bristol stool chart) on test day +1
Stool consistency+2 | 48hr
  Stool consistency (Bristol stool chart) on test day +2
Abdominal pain-3 | -72hr
  Abdominal pain (Likert scale 0-10) on test day -3
Abdominal pain-2 | -48hr
  Abdominal pain (Likert scale 0-10) on test day -2
Abdominal pain-1 | -24hr
  Abdominal pain (Likert scale 0-10) on test day -1
Abdominal pain-T | Testday (0hr)
  Abdominal pain (Likert scale 0-10) on test day
Abdominal pain+1 | 24hr
  Abdominal pain (Likert scale 0-10) on test day +1
Abdominal pain+2 | 48hr
  Abdominal pain (Likert scale 0-10) on test day +2
Bloating-3 | -72hr
  Bloating (Likert scale 0-10) on test day -3
Bloating-2 | -48hr
  Bloating (Likert scale 0-10) on test day -2
Bloating-1 | -24hr
  Bloating (Likert scale 0-10) on test day -1
Bloating-T | Testday (0hr)
  Bloating (Likert scale 0-10) on test day
Bloating+1 | 24hr
  Bloating (Likert scale 0-10) on test day +1
Bloating+2 | 48hr
  Bloating (Likert scale 0-10) on test day +2
Flatulence-3 | -72hr
  Flatulence (Likert scale 0-10) on test day -3
Flatulence-2 | -48hr
  Flatulence (Likert scale 0-10) on test day -2
Flatulence-1 | -24hr
  Flatulence (Likert scale 0-10) on test day -1
Flatulence-T | Testday (0hr)
  Flatulence (Likert scale 0-10) on test day
Flatulence+1 | 24hr
  Flatulence (Likert scale 0-10) on test day +1
Flatulence+2 | 48hr
  Flatulence (Likert scale 0-10) on test day +2
Nausea-3 | -72hr
  Nausea (Likert scale 0-10) on test day -3
Nausea-2 | -48hr
  Nausea (Likert scale 0-10) on test day -2
Nausea-1 | -24hr
  Nausea (Likert scale 0-10) on test day -1
Nausea-T | Testday (0hr)
  Nausea (Likert scale 0-10) on test day
Nausea+1 | 24hr
  Nausea (Likert scale 0-10) on test day +1
Nausea+2 | 48hr
  Nausea (Likert scale 0-10) on test day +2
Heartburn-3 | -72hr
  Heartburn (Likert scale 0-10) on test day -3
Heartburn-2 | -48hr
  Heartburn (Likert scale 0-10) on test day -2
Heartburn-1 | -24hr
  Heartburn (Likert scale 0-10) on test day -1
Heartburn | Testday (0hr)
  Heartburn (Likert scale 0-10) on test day
Heartburn+1 | 24hr
  Heartburn (Likert scale 0-10) on test day +1
Heartburn+2 | 48hr
  Heartburn (Likert scale 0-10) on test day +2

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No